CLINICAL TRIAL: NCT05102409
Title: An Exploratory, Single-Center, Double-Masked, Crossover Clinical Trial to Assess Safety and Tolerability of 0.25% Reproxalap Ophthalmic Solution Compared to Xiidra® in Subjects With Dry Eye Disease in a Dry Eye Chamber
Brief Title: An Exploratory Crossover Clinical Trial to Compare the Activity of Reproxalap and Lifitegrast in a Dry Eye Disease Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-025
Record Dates: First submitted 2021-10-18; First posted 2021-11-01 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2021-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental): Single dose
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Xiidra® (5% lifitegrast ophthalmic solution) (Active Comparator): Single dose
  Interventions: Drug: Xiidra® (5% lifitegrast ophthalmic solution)

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) dosed once
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Xiidra® (5% lifitegrast ophthalmic solution) — Xiidra® (5% lifitegrast ophthalmic solution) dosed once
  Arms: Xiidra® (5% lifitegrast ophthalmic solution)

SUMMARY:
An Exploratory, Single-Center, Double-Masked, Crossover Clinical Trial to Assess Safety and Tolerability of 0.25% Reproxalap Ophthalmic Solution Compared to Xiidra® in Subjects with Dry Eye Disease in a Dry Eye Chamber

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen (18) to70 years of age at the time of screening (either gender and any race).
2. Ability to provide written informed consent.
3. Reported history of dry eye for at least 6 months prior to Visit 1.

Exclusion Criteria:

1. Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal) or active ocular inflammation at Visit 1.
2. Contact lens use within 7 days of Visit 1 or anticipate using contact lenses during the trial.
3. A condition that the investigator feels may put the subject at significant risk may confound the study results or may interfere significantly with the subject's participation in the trial.
4. Inability or unwillingness to follow instructions, including participation in all study assessments/procedures and visits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-six subjects were enrolled in a two-period crossover design trial in which each subject received lifitegrast and reproxalp during separate treatment periods separated by approximately 7 days. Subjects were dosed once for each treatment period just before entry into a 45-minute dry eye chamber.
Groups:
- Lifitegrast, Reproxalap: Subjects received a single dose of 5% lifitegrast ophthalmic solution just before dry eye chamber entry, followed by a seven-day washout. Subjects then received a single dose of 0.25% reproxalap just before dry eye chamber entry.
Period: Overall Study
Arm/Group | Lifitegrast, Reproxalap
Started | 56
Completed | 54
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Enrolled subjects
Arm/Group | Lifitegrast, Reproxalap
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 33
  More than one race | 5
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Discomfort
Description: Ocular discomfort (0 = none, 10 = extremely severe) was reported by patients in a dry eye chamber. Change from baseline was analyzed using a mixed model repeated measures (MMRM) analysis, with baseline as a covariate, and treatment and intra-chamber time point as factors.
Time Frame: The efficacy assessment period was approximately every 5 minutes during a 45-minute dry eye chamber. Baseline was prior to dosing for each treatment period.
Population: Safety population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Reproxalap: Reproxalap dosed topically prior to dry eye chamber entry
- Lifitegrast: Lifitegrast dosed topically prior to dry eye chamber entry
Arm/Group | Reproxalap | Lifitegrast
Number analyzed (Participants) | 54 | 56
score on a scale | 1.35 (0.21) | 2.07 (0.25)

2. Primary Outcome: Change From Baseline in Ocular Itching
Description: Ocular itching (0 = none, 10 = extremely severe) was reported by patients in a dry eye chamber. Change from baseline was analyzed using a MMRM analysis, with baseline as a covariate, and treatment and intra-chamber time point as factors.
Time Frame: as for outcome 1
Population: Safety population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Reproxalap | Lifitegrast
Number analyzed (Participants) | 54 | 56
score on a scale | 0.93 (0.21) | 1.54 (0.25)

ADVERSE EVENTS:
Time Frame: One day for each intervention
Arm/Group | Reproxalap | Lifitegrast
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 40/54 | 12/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reproxalap (N=54) | Lifitegrast (N=56)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 6 (6)
General Disorders (General disorders) | 40 (40) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT05102409/Prot_SAP_001.pdf